CLINICAL TRIAL: NCT06255119
Title: The Feasibility of 3D Therapy Thrive for Inpatients With Opioid Use Disorder
Brief Title: The Feasibility of VR for OUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3D Therapy, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 2022/03/9
Record Dates: First submitted 2023-06-20; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-10

CONDITIONS: Opioid Use Disorder
Keywords: mood; cravings; retention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects were blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active VR Group (Active Comparator): Participants received the active virtual therapy intervention.
  Interventions: Device: 3D Therapy Thrive
- Control Group (No Intervention): A group of patients concurrently on the ATS unit, otherwise eligible to participate in the study who did not enroll, and did not receive an intervention.

INTERVENTIONS:
Device: 3D Therapy Thrive — A novel virtual reality software intervention that utilizes elements of Cognitive Behavioral Therapy to improve outcomes for inpatients with OUD.
  Arms: Active VR Group

SUMMARY:
This study aims to evaluate feasibility of a virtual reality software device and measure the effects of the intervention on OUD patient mood, tension and cravings, as well as the effect of treatment on patient retention to their inpatient detox protocol.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility and preliminary effectiveness of a novel virtual reality (VR) based intervention; 3D Therapy Thrive (3DTT). Inpatient detoxification can improve outcomes for individuals with opioid use disorder (OUD), however patients often leave treatment early due to mood, tension, and cravings associated with opioid withdrawal. Subjects were recruited from a community inpatient detoxification program and received up to two sessions of 3DTT. The patients completed surveys to assess their mood, distress, cravings, and overall satisfaction with the experience. Retention was measured by protocol completion as reported by clinic staff, independent of the study. A group of patients with OUD consecutively admitted to the program comprised a comparison treatment-as-usual (TAU) group.

ELIGIBILITY:
Inclusion Criteria

1.18 years or older

2. Current diagnosis of opioid use disorder

3. Current inpatient in detox ATS unit

4. Fluent in English

Exclusion Criteria

1. Active suicidality
2. History of seizures
3. History of psychosis
4. Severe visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Retention in Treatment | At departure from facility, through study completion, an average of 10 days
  Medical record indicating whether patient completed detox protocol (i.e., completed, left against medical advice, administratively discharged, or moved to higher level of care)
Feasibility and Tolerability of 3DTT | Immediately after each treatment
  Feasibility and tolerability of 3DTT was measured by the Side Effects Questionnaire.

SECONDARY OUTCOMES:
Mood | Before and after each treatment, approximately every other day for up to 5 days
  Depressive symptoms as measured by the AB-POMS depression scale (0-4, not at all to extremely)
Anxiety | Before and after each treatment, approximately every other day for up to 5 days
  Anxiety symptoms as measured by the AB-POMS scale (0-4, not at all to extremely)
Cravings | Before and after each treatment, approximately every other day for up to 5 days
  Opioid cravings as measured by the Visual Analog Scale (1-10, with higher scores indicating greater cravings.)

CONTACTS AND LOCATIONS:
Locations (1):
- The Gavin Foundation, Quincy, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No